CLINICAL TRIAL: NCT07051421
Title: A NEW EARLY WARNING SCORE TO SUPPORT CLINICAL DECISION PROCESSES IN POSTANESTHETIC FOLLOW-UP: RECO-EWS
Brief Title: RECOVERY ROOM EARLY WARNING SCORE
Status: Not yet recruiting | Type: Observational
Sponsor: Istinye University (Other)
Responsible Party: Principal Investigator, İlke Dolgun, ASSOC.PROF., Haseki Training and Research Hospital
Other Study IDs: HASEKI AHMET TEZ
Record Dates: First submitted 2025-06-26; First posted 2025-07-04 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-06

CONDITIONS: Early Warning Score
MeSH Terms: interventions — Early Warning Score

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: EARLY WARNING SCORE — In the RECO-EWS scoring system we designed; 0-7 low risk, 7-10 medium risk, ≥10 high risk, postoperative stay findings of high-risk patients and, if necessary, new cut-off values are determined for each parameter in the scoring system according to the analysis results.

SUMMARY:
In this study, we aimed to develop a scoring system that facilitates patient risk stratification in the recovery room during the postanesthetic follow-up period and can objectively identify patients in need of early intervention.

ELIGIBILITY:
Inclusion Criteria:

* Those over 18 years of age,
* Those in ASA I-III class,
* Those who have undergone planned elective surgery under general anesthesia,
* Those who have been informed about the study in advance and given their consent.

Exclusion Criteria:

* Those under 18 years of age,
* Those who underwent emergency intervention,
* Those in the ASA-Ⅳ class,
* Those who underwent regional anesthesia,
* Those with a history of cognitive retardation, visual-hearing impairment or psychiatric disease that prevents communication, those who have previously been diagnosed with neurocognitive disorders,
* Patients who could not complete the procedure, patients with data loss,
* Patients whose general anesthesia duration is less than 90 minutes will not be included in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over 18 years of age, in ASA class I-III, who have undergone planned elective surgery under general anesthesia, and who have been informed and given informed consent in advance of the study.
Sampling Method: Non-Probability Sample
Enrollment: 208 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
RECO-EWS | 24 HOURS
  0-7 low risk, 7-10 medium risk, ≥10 high risk

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Pazar B, Yava A. Evaluation of Early Warning Scoring System and Nursing Guide Application in Post-Anaesthesia Care Unit. Turk J Anaesthesiol Reanim. 2013 Dec;41(6):216-22. doi: 10.5152/TJAR.2013.37. Epub 2013 May 23. PMID 27366375
- [Result] Mert S, Kersu O, Cesur S, Topbas O, Erdogan S. The Effect of Modified Early Warning Score (MEWS) and Nursing Guide Application on Postoperative Patient Outcomes: A Randomized Controlled Study. J Perianesth Nurs. 2024 Aug;39(4):596-603. doi: 10.1016/j.jopan.2023.10.023. Epub 2024 Feb 1. PMID 38300197